CLINICAL TRIAL: NCT05092503
Title: A Phase I/Ⅱ Randomized Controlled Proof-of-concept Study to Evaluate the Safety and Efficacy of JINZHEN Granules for Oral Solution in Participants With Mild to Moderate COVID-19
Brief Title: JINZHEN for Treatment of Mild to Moderate COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lianyungang Kanion Group, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JZ-2001-01
Record Dates: First submitted 2021-10-06; First posted 2021-10-25 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- JINZHEN low dose arm (Experimental): Patients will take 0.375 gram of JINZHEN Granules twice a day for 14 days.
  Interventions: Drug: JINZHEN Granules for Oral Solution
- JINZHEN middle dose arm (Experimental): Patients will take 0.75 gram of JINZHEN Granules twice a day for 14 days.
  Interventions: Drug: JINZHEN Granules for Oral Solution
- JINZHEN high dose arm (Experimental): Patients will take 1.5 gram of JINZHEN Granules twice a day for 14 days.
  Interventions: Drug: JINZHEN Granules for Oral Solution
- Placebo arm (Placebo Comparator): Patients will take placebo granules twice a day for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JINZHEN Granules for Oral Solution — JINZHEN granules will be dissolved in drinking water and administered orally.
  Arms: JINZHEN high dose arm; JINZHEN low dose arm; JINZHEN middle dose arm
Drug: Placebo — Placebo granules will be dissolved in drinking water and administered orally.
  Arms: Placebo arm

SUMMARY:
JINZHEN is a botanical drug that contains eight chemical constituents extracted from plant, mineral and animal origin raw materials. This study is to evaluate the safety and efficacy of JINZHEN Granules for Oral Solution compared to placebo for treatment of mild to moderate COVID-19 outpatients.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, placebo-controlled, proof of concept study with four groups (low dose treatment group, middle dose treatment group, high dose treatment group, and placebo group). Study eligibility will be assessed during screening. Study participants will be randomized in a 3:1 ratio to receive JINZHEN Granules for Oral Solution or placebo granules for 14 days.

During the 14-day clinical study, participants will be assessed daily at home using e-diary to collect clinical data and in person visit on Day 7 and Day14. All subjects will undergo a series of efficacy, safety, and laboratory assessments. Clinical observation endpoints will be assessed at day 7 and day 14. Interim analysis will be performed to evaluate efficacy and safety of 7-day and 14-day treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 years and ≤ 50 years of age, BMI < 30 at time of enrollment.
2. Have presence of SARS-CoV-2 infection confirmed by reverse transcription polymerase chain reaction (RT-PCR) test with sample collection ≤ 3 days prior to randomization.
3. Fever ≥ 38.0℃ (100.4℉ oral temperature) or ≥ 38.6℃ (101.48℉ tympanic temperature) within 48 hours before screening; and at least one of respiratory rate > 24 breaths/minute or cough (scored ≥ 2 via participant questionnaire).
4. Initial onset of signs/symptoms for ≤ 5 days prior to randomization.
5. Participant provides written informed consent prior to initiation of any study procedures.
6. Participant is willing to accept randomization to any assigned treatment arm. And participant understands and agrees to comply with planned study procedures.

Exclusion Criteria:

1. SARS-CoV-2 infection confirmed participants who are currently hospitalized or are expected to need hospitalization (for COVID-19 within 48 hours of randomization).
2. Participants who have SpO2 ˂ 93% on room air at sea level, or respiratory frequency ˃ 30 breaths/minute, or heart rate ≥ 125 per minute.
3. Require mechanical ventilation or anticipated impending need for mechanical ventilation.
4. Pre-existing pulmonary conditions such as chronic obstructive pulmonary disease or asthma. Imaging confirmed the existence of severe lung interstitial lesions, bronchiectasis, bronchopulmonary dysplasia and other basic pulmonary diseases. Have chronic pulmonary diseases such as pulmonary embolism and pulmonary hypertension at present.
5. Have any other active infectious diseases. Such as influenza, bacterial infections of the respiratory system (suppurative tonsillitis, acute tracheobronchitis, active tuberculosis, etc.) and other respiratory diseases affecting the evaluation of clinical trials.
6. ALT/AST > 3×ULN, TBIL ≥ 1.5×ULN, creatinine ≥ 1.5×ULN.
7. Patients with recurrent diarrhea or abnormal intestinal function that are not caused by COVID-19.
8. Patients with a history of type 1 or type 2 diabetes, OR with glycosylated hemoglobin (HbA1c) level ≥ 6.5% during screening.
9. Patients with hypertension at screening (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg).
10. Have any serious concomitant systemic disease, condition or disorder that, in the opinion of the investigator, should preclude participation in this study. Such as, unresectable malignant tumor, blood disease, active bleeding, cachexia, nervous system disease, endocrine system disease, cardiovascular disease and heart conditions (e.g., heart failure [New York heart association (NYHA) ≥ grade 3], coronary artery disease, cardiomyopathies), down syndrome, sickle cell disease, cystic fibrosis, thalassemia, etc.
11. Suffering from diseases that seriously affect the immune system, such as HIV infection, splenectomy, organ or blood stem cell transplantation, etc.
12. Participants who received systemic corticosteroids or other immunosuppressive medications within 14 days before screening.
13. Participants with positive results of hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) at screening period.
14. Participants who are using any herb supplements/products.
15. Participants who are currently using anti-virus drugs.
16. Nursing women or women of pregnancy test positive or planning to be pregnant throughout the study period.
17. Psychiatric or cognitive illness (such as schizophrenia spectrum disorders, mood disorders, dementia, etc.) or alcohol abuse.
18. Participants who have received any interventional experimental treatment for COVID-19 within the 30 days prior to the time of the screening evaluation.
19. Participants unable to take oral medications.
20. Participants who plan to receive live attenuated vaccine within 1 month prior to the first administration of the study drug or during the study period.
21. Participants with mild to moderate COVID-19 who would be eligible for another FDA authorized COVID-19 therapeutic.
22. Participants who are on sensitive substrates or substrates of a narrow therapeutic range for major cytochrome P450 and transporters.
23. Other conditions inappropriate for participation in this clinical trial considered by the investigators.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Median time to sustained symptom resolution within 28 days after beginning of administration. | 28 days
  * Sustained symptom resolution is defined as absences of symptoms (except for mild fatigue or mild cough) over at least 2 days.
  * Time to sustained symptom resolution is defined as the time from initiation of study treatment (active or placebo) until symptom resolution.

SECONDARY OUTCOMES:
Proportion of participants who experience any of these events within 14 and 28 days after beginning of administration. | up to Day 14 and 28
  COVID-19 related hospitalization (defined as > 24 hours of acute care).
  COVID-19 related emergency room visit > 24 hours.
  All-cause mortality.
Proportion of participants with clinical recovery of symptomatic reliefs within 7 days and 14 days after beginning of administration. | up to Day 7 and 14
  Clinical recovery is defined as subjects with normalization of fever, respiratory rate, and oxygen saturation, and alleviation of cough, sustained for at least 2 days.
Proportion of participants demonstrating improvement of each targeted symptom via participant questionnaire. | up to Day 7, 14 and 28
  Improvement is defined as symptoms scored 2 or 3 at baseline are scored 0 or 1, AND symptoms scored 1 at baseline are scored 0.
Proportion of participants demonstrating resolution of each targeted symptom via participant questionnaire. | up to Day 7, 14 and 28
  Resolution is defined as symptoms (except tiredness and cough) scored ≥ 1 at baseline are scored 0, AND tiredness or cough scored > 1 at baseline are scored ≤ 1.
Time to Clinical Recovery (TTCR). | up to Day 7 and 14
  TTCR is defined as the time from initiation of study treatment (active or placebo) until clinical recovery.
Time to improvement of each targeted symptom via participant questionnaire. | up to Day 7, 14 and 28
  Time to improvement is defined as the time from initiation of study treatment (active or placebo) until this symptom meets the definition of improvement AND sustained for at least 2 days.
Time to resolution of each targeted symptom via participant questionnaire. | up to Day 7, 14 and 28
  Time to resolution is defined as the time from initiation of study treatment (active or placebo) until this symptom meets the definition of resolution AND sustained for at least 2 days.
Viral load change | Day 8 and 15
  Viral load change from screening to Day 8 and 15

CONTACTS AND LOCATIONS:
Overall Officials: Zhu, Study Director — Jiangsu Kanion Pharmaceutical Co., Ltd
Locations (10):
- United States (10):
  - Clearview Medical Research LLC, Canyon Country, California
  - Family First Medical Research Center, Hialeah Gardens, Florida
  - LMG Research, Miami, Florida
  - AA Medical Research Center, Flint, Michigan
  - F. Gabriel LLC, Bayonne, New Jersey
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - Frontier Clinical Research LLC, Smithfield, Pennsylvania
  - Piedmont Research Partners, Fort Mill, South Carolina
  - SMS Clinical Research, Mesquite, Texas
  - Frontier Clinical Research LLC, Morgantown, West Virginia